CLINICAL TRIAL: NCT00611312
Title: Effects of Intense Cognitive Training on Standardized Measures of Cognition in Those With Very Mild Alzheimer's Disease
Brief Title: Effects of Delivery Mode of Cognition Intervention in Early Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Yvonne Colgrove, PT, PhD, Principal Investigator, University of Kansas
Organization: University of Kansas Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IIRG-07-57789; 11008
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; Cognitive training
MeSH Terms: conditions — Alzheimer Disease | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Cognitive Training
  Interventions: Behavioral: Cognitive Training

INTERVENTIONS:
Behavioral: Cognitive Training — Intense cognitive training, two consecutive weeks, each weekday, 6 hours/day

SUMMARY:
The purpose of this study is to see if an intense two-week long cognitive training program helps the thinking ability of adults with very mild Alzheimer Disease. We anticipate that scores on clinical cognitive tests will be better after the training.

DETAILED DESCRIPTION:
Twenty of the 30 subjects will be recruited to participate in functional magnetic resonance imaging (fMRI). Scanning will be done while subjects perform a verbal learning task. Ten subjects will be scanned before and after the two week training. Another ten will be scanned twice at a two week interval before beginning the cognitive training.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of very mild Alzheimer's Disease (CDC of 0.5) and mild Alzheimer's Disease (CDC of 1.0)

Exclusion Criteria:

* Neurologic disorder other than Alzheimer's disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-02; Primary Completion 2012-05 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Composite score of 5 cognitive tests including 1)WAIS digit span, 2) word fluency, 3) trail making test-A 4) Rey Osterrieth complex figure and 5) MMSE | 2 weeks with FU at 2 and 4 months

SECONDARY OUTCOMES:
Brain activity during functional brain imaging | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Colgrove, PhD, PT, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States